CLINICAL TRIAL: NCT02835014
Title: Mental Health Screenings in Adolescents With Type I Diabetes
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L16-118
Record Dates: First submitted 2016-07-05; First posted 2016-07-15 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus Type I
Keywords: Diabetes Mellitus Type I; Adolescents; Mental Health; Self efficacy; parenting styles
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adolescents with T1DM: Adolescents with type I Diabetes Mellitus diagnosed for at least one year will be screened for mental health symptoms with the PHQ9, SCARED and UCLA PTSD. Self-efficacy regarding self-care and diabetes management will be assessed by using the SEDM. Parenting styles will be assessed by administering the Parenting Styles and Dimensions Questionnaire (PSDQ).
  Interventions: Behavioral: Mental Health Symptoms; Behavioral: Self-efficacy regarding self-care and diabetes management; Behavioral: Parenting Styles

INTERVENTIONS:
Behavioral: Mental Health Symptoms — Adolescents with T1DM will be asked to complete PHQ9 (depression screening), SCARED (anxiety screening) and UCLA PTSD (trauma screening)
  Other Names: PHQ9; SCARED; UCLA PTSD
Behavioral: Self-efficacy regarding self-care and diabetes management — Adolescents with T1DM will be asked to complete the SEDM to asses self-efficacy for diabetes management
  Other Names: SEDM
Behavioral: Parenting Styles — Parents of adolescents with T1DM will be asked to complete the PSDQ to asses parenting style
  Other Names: Parenting Styles and Dimensions Questionnaire (PSDQ)

SUMMARY:
This study will focus on screening for mental health symptoms in adolescents with type 1 diabetes mellitus (T1DM) while assessing the relationship of these symptoms with a parent-reported parenting styles survey, and the youth's report of their ability to manage their own diabetes care through a self-efficacy survey. Gender differences will be explored in relation to the different measures.

DETAILED DESCRIPTION:
Background: More than 200,000 youth in the United States are affected by T1DM, a chronic illness that results from an absolute insulin secretion deficiency. Like other chronic illnesses, T1DM is a known risk factor for additional health related comorbidities. Furthermore, parenting this particular group of adolescents can present its own unique challenges and earlier research has established that parenting styles undoubtedly influence a child's ability to manage their own care and metabolic control. Although mental health disorders are common among adolescents, diabetic youth are reported to be at even higher risk for mental health symptoms and adjustment issues. Often, after a diagnosis of T1DM adolescent youth may develop anxiety, sadness, and experience social withdrawal. In fact, ∼30% of children develop a clinical adjustment disorder within the first 3 months post diagnosis. However, these early struggles often resolve within the first year; nevertheless, poor adaptation during the initial maladjustment phase has shown to be indicative of later mental health symptoms. The risk of suicide or suicide ideation in patients with T1DM is prevalent. Previous studies have found that girls with type 1 diabetes appear to be more affected with depression, and anxiety than are boys with type 1 diabetes. Additionally, adolescent females are at a higher risk of presenting with recurrent diabetic ketoacidosis (DKA) than adolescent males. It has also been established that maladaptive child responses to an acute or chronic medical condition can result in stress symptoms. Despite T1DM's classification as a treatable or manageable illness, failing to adhere to the prescribed treatment regimen can have catastrophic results. Severe outcomes can include blindness, DKA, coma, and even death. The mere daily threat of experiencing one of these conditions can be enough to evoke a traumatic response. Although there is a plethora of studies reporting clinically significant rates of post traumatic stress disorder (PTSD) in children who have experienced traumatic injuries, transplants, and even cancer, fewer studies have aimed at assessing post-traumatic stress responses to T1DM. Self-Efficacy is defined as the belief that one can be successful in completing a specific task in a given situation. Adolescent ability to self-manage a chronic illness can be negatively impacted by mental health comorbidities. More specifically, these mental health comorbidities correlate to poor glycemic control. Previous studies investigating Self-Efficacy in adolescents solidified the connection of Self-Efficacy to diabetes mellitus and glycemic control. Positive and adequate parental involvement for diabetes care is consistently associated with improved metabolic control and adherence. Adolescence is marked as a time for increased autonomy, privacy and responsibility, so constructing a dynamic balance that includes parental involvement and support to ensure proper daily T1DM care seems an ever present challenge. Parenting style may be a more specific predictor for diabetes outcomes than other contextual aspects related to the family since youth with type 1 diabetes typically depend on their parents' help when managing the condition. Three categories of parenting styles have been described, Authoritarian, Permissive and Authoritative. Authoritarian parents have high level of assertiveness and control in their implementation of structure and clear definitions of rules but express very low levels of responsiveness. Alternatively, permissive parents are typically associated with addressing childrens' emotional needs yet provide little structure or guidance through boundaries. Authoritative parents fall between authoritarian and permissive by maintaining a strong but appropriate structure and nurturing amounts of responsiveness and warmth. Research has shown parental style to directly affect a child's health outcome, specifically, authoritative parenting behaviors are associated with positive health outcomes including better glycemic index control, improved adolescent self-care practices, and well-being with regards to internalizing and externalizing behaviors. Previous literature has identified connections between gender, parenting style, and mental illness. For example, females have shown to be more responsive to parenting style as exemplified through increased occurrences of depression and poorer adherence when the adolescents view the mother as controlling. The relational component exhibited through this trend could indicate a vulnerability, more present in girls than boys, considering the interpersonal dynamic between parent and child associated with parenting style.

This study will examine whether or not adolescent girls from New Mexico and West Texas diagnosed with T1DM longer than one year are more likely to be affected with mental health issues than their male counterparts and to ascertain the impact of these issues on glycemic control. Participants will be screened for mental health symptoms using three brief instruments currently used in general practice. Additionally, youth reported self-efficacy and parenting styles will be assessed. The identified instruments are widely used in pediatric clinical and research settings and are appropriate for this age group. Upon completion of each screening the appropriate follow up care or referral for services will be completed in the interest of patient care. A chart review will be conducted at enrollment to obtain demographic information and a history of diabetes management and care, then again at 12 months after the enrollment.

Significance: This will be the first study to screen for depression, anxiety, and trauma mental health symptoms in youth with T1DM within the west Texas - eastern New Mexico geographic region served by Texas Tech University Health Sciences Center (TTUHSC). Additionally, self-reported parenting behaviors and parenting styles will be identified. Gender and racial differences among the participants will be analyzed with respect to parent reported parenting style. The robust Latino population, combined with the rural community setting provides a unique perspective regarding measured outcomes. Furthermore, amidst the wave of implementation of trauma-informed care services across the United States, the field calls for a closer look at the traumatic experiences resulting from type I diabetes complications, many of which can be life threatening, and have been found to lead to traumatic stress symptomatology. The data collected in this study may serve to inform future directions regarding screening protocols and interventions created to address these issues and subsequently impact diabetes control and complications among this population.

Aim: This study aims to assess mental health symptoms and self-efficacy in youth with T1DM receiving care in the TTUHSC pediatric endocrine clinic. Furthermore the study seeks to analyze the relationships among mental health, parent-reported parenting styles and youth-reported self-efficacy regarding self-care and diabetes management. Gender and racial differences will be discussed.

Hypotheses: Adolescent females are more likely to be affected with mental health symptoms than their male counterparts. Positive mental health screens will be associated with lower self-efficacy regardless of parenting style. Authoritative style parenting will be associated with higher self-efficacy, fewer positive mental health screenings, and encounters of diabetes complications. Authoritative style parenting will be positively associated with diabetes control. Authoritarian style parenting will be associated with lower self-efficacy, positive mental health screenings. Authoritarian and permissive style parenting will be associated with poor diabetes control, and encounters of diabetes complications. Lastly, those who seek mental health services will see improvement with diabetes control (defined by hemoglobin A1C levels equal or less than 8.5%) and will be less likely to present to the emergency room, require hospital admission due to DKA or other complications of T1DM.

Study Design and Methods: On May 17th, 2016 the study received IRB approval. Once the trial gets registered on ClinicalTrials.Gov, participants will be recruited for enrollment into the study.

Procedures: 1) Study Coordinator will be notified of potential study participants presenting to the pediatric endocrine clinic. 2) If the patient meets inclusion criteria for the study, the coordinator will ask for consent/assent to participate. 3) Demographic Information will be obtained: age at diabetes diagnosis, number of year since diagnosis, gender, zip code, race/ethnicity, maternal education, insurance type, length of residence at current home, anticipated housing relocation, length of employment at current job, anticipated parental job changes, previous mental health screenings and interventions, number of previous DKA episodes per year, diabetes control over time by looking at HbA1C measurements during admissions to the hospital or during office follow up. 4) Mental Health Screen/Assessment - Study participants will be screened for mental health symptoms using the following screening instruments: Patient Health Questionnaire for Depression (PHQ - 9), Screen for Child Anxiety Related Emotional Disorders (SCARED), University of California Los Angeles (UCLA PTSD) Reaction Index - abbreviated version, Youth participants will also complete the Self-Efficacy for Diabetes Self-Management scale (SEDM), a parent will complete the self-reported Parenting Styles and Dimensions Questionnaire (PSDQ). 5) Follow Up to Assessment: If patient indicates thoughts of self-harm or suicide ideation on question 9 of the PHQ-9, then the C-SSRS Screener version with triage points risk assessment will be conducted to determine if Emergency room follow up is necessary. Actively suicidal patients will be referred to the emergency room (ER) for immediate evaluation as per standard of care. Those non suicidal patients but with a positive mental health screening(s) will be provided with referral and resource information including a list of mental health providers if desired. 6) Initial data will be entered and de-identified in the data base, hard copies will be kept in order to properly match the participants after the chart review. 7) Twelve months after the initial mental health screening a chart review will be conducted to collect the following information: Hemoglobin A1C levels in the preceding 12 months ii, number of follow up visits with pediatric endocrinology, number of ER visits, number of hospital admissions, number of DKA episodes, suicidal Ideation or suicidal Attempts (SA), Non-Suicidal self-injury (NSSI), number of visits to mental health providers (If unable to obtain this information through their medical chart, then individual mental health providers-from the list provided on initial screening - will be contacted to obtain the number of visits during the preceding 12 months). Data will be entered and de-identified for analysis. At this time any hard copies of the assessments will be destroyed.

Statistical Analysis: All demographic data will be expressed as mean + SD and frequencies (%). The differences between males and females will be analyzed using the Student's t-test for continuous data and with Chi Square for categorical data during the initial analysis. A two-tailed p value of <0.05 will be considered statistically significant. Additional analyses will include ANOVA or MANOVA or a regression model during the full analysis. The latest SPSS software version will used for statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients' from west Texas or eastern New Mexico ages 12-17 years old, who have been diagnosed with Type I diabetes for at least one year from the time of enrollment, who present to the pediatric endocrine clinic for care.

Exclusion Criteria:

* Patients who are younger than 12 years old or older than 17 years old. Patients who were diagnosed less than one-year ago from time of recruitment will also be excluded. Or, those who decline to participate.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents from West Texas or Eastern New Mexico ages 12-17 years old diagnosed with type I diabetes for at least one year from the time of enrollment presenting to the pediatric endocrine clinic at Texas Tech University Health Sciences Center for care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with a positive depression screening | Available immediately after scoring patient's PHQ9 questionnaire
  The PHQ9 questionnaire will be used to identify those patients with depression symptoms, and the total score will allow us to grade the depression into minimal, mild, moderate, moderately severe or severe. At the end of recruitment period we will be able to compare results by gender as well.

SECONDARY OUTCOMES:
Number of patients with a positive anxiety screening | Available immediately after scoring patient's SCARED questionnaire
  The SCARED questionnaire will be used to identify those patients with anxiety symptoms for those scoring greater than 25, as well as to identify those with different categories of anxiety such as panic disorder, generalized anxiety disorder, social anxiety, separation anxiety and school avoidance by using the cut off values provided on the screening questionnaire for each category. At the end of recruitment period we will be able to compare results by gender as well
Number of patients with positive PTSD | Available immediately after scoring patient's UCLA PTSD questionnaire
  The UCLA PTSD questionnaire will be used to identify those patients with PTSD symptoms as well as the severity based on total score
Improvement in Diabetes Control defined by HbA1C equal or lower than 8.5% | One year after screenings were administered and referrals were suggested

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Nur, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Craig ME, Hattersley A, Donaghue KC. Definition, epidemiology and classification of diabetes in children and adolescents. Pediatr Diabetes. 2009 Sep;10 Suppl 12:3-12. doi: 10.1111/j.1399-5448.2009.00568.x. No abstract available. PMID 19754613
- [Background] Silverstein J, Klingensmith G, Copeland K, Plotnick L, Kaufman F, Laffel L, Deeb L, Grey M, Anderson B, Holzmeister LA, Clark N; American Diabetes Association. Care of children and adolescents with type 1 diabetes: a statement of the American Diabetes Association. Diabetes Care. 2005 Jan;28(1):186-212. doi: 10.2337/diacare.28.1.186. No abstract available. PMID 15616254
- [Background] Mlynarczyk SM. Adolescents' perspectives of parental practices influence diabetic adherence and quality of life. Pediatr Nurs. 2013 Jul-Aug;39(4):181-9. PMID 24027952
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Cameron FJ, Northam EA, Ambler GR, Daneman D. Routine psychological screening in youth with type 1 diabetes and their parents: a notion whose time has come? Diabetes Care. 2007 Oct;30(10):2716-24. doi: 10.2337/dc07-0603. Epub 2007 Jul 20. No abstract available. PMID 17644619
- [Background] Corathers SD, Kichler J, Jones NH, Houchen A, Jolly M, Morwessel N, Crawford P, Dolan LM, Hood KK. Improving depression screening for adolescents with type 1 diabetes. Pediatrics. 2013 Nov;132(5):e1395-402. doi: 10.1542/peds.2013-0681. Epub 2013 Oct 14. PMID 24127480
- [Background] Naar-King S, Podolski CL, Ellis DA, Frey MA, Templin T. Social ecological model of illness management in high-risk youths with type 1 diabetes. J Consult Clin Psychol. 2006 Aug;74(4):785-9. doi: 10.1037/0022-006X.74.4.785. PMID 16881786
- [Background] Kovacs M, Iyengar S, Goldston D, Stewart J, Obrosky DS, Marsh J. Psychological functioning of children with insulin-dependent diabetes mellitus: a longitudinal study. J Pediatr Psychol. 1990 Oct;15(5):619-32. doi: 10.1093/jpepsy/15.5.619. PMID 2283571
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Schwartz DD, Cline VD, Axelrad ME, Anderson BJ. Feasibility, acceptability, and predictive validity of a psychosocial screening program for children and youth newly diagnosed with type 1 diabetes. Diabetes Care. 2011 Feb;34(2):326-31. doi: 10.2337/dc10-1553. Epub 2011 Jan 7. PMID 21216856
- [Background] Pompili M, Forte A, Lester D, Erbuto D, Rovedi F, Innamorati M, Amore M, Girardi P. Suicide risk in type 1 diabetes mellitus: A systematic review. J Psychosom Res. 2014 May;76(5):352-60. doi: 10.1016/j.jpsychores.2014.02.009. Epub 2014 Feb 28. PMID 24745775
- [Background] Roy A, Roy M, Janal M. Suicide attempts and ideation in African-American type 1 diabetic patients. Psychiatry Res. 2010 Aug 30;179(1):53-6. doi: 10.1016/j.psychres.2010.06.004. Epub 2010 Jul 13. PMID 20630602
- [Background] de Wit M, Snoek FJ. Depressive symptoms and unmet psychological needs of Dutch youth with type 1 diabetes: results of a web-survey. Pediatr Diabetes. 2011 May;12(3 Pt 1):172-6. doi: 10.1111/j.1399-5448.2010.00673.x. PMID 20561242
- [Background] Rewers A, Chase HP, Mackenzie T, Walravens P, Roback M, Rewers M, Hamman RF, Klingensmith G. Predictors of acute complications in children with type 1 diabetes. JAMA. 2002 May 15;287(19):2511-8. doi: 10.1001/jama.287.19.2511. PMID 12020331
- [Background] Pollin, I., (1995). Medical crisis counseling: Short-term therapy for long-term illness. New York: W.W. Norton.
- [Background] Bronfman, E. T., Biron Campis, L., & Koocher, G. P. (1998). Helping children to cope: Clinical issues for acutely injured and medically traumatized children. Professional Psychology: Research and Practice, 29(6), 574.
- [Background] Karczewski, S. A. (2015). Pediatric Medical Traumatic Stress in Youth with Type 1 Diabetes and Their Caregivers: A Longitudinal Assessment of Metabolic Control and Psychosocial Mediators (doctoral dissertation). DePaul University, Chicago, IL.
- [Background] Bruce M. A systematic and conceptual review of posttraumatic stress in childhood cancer survivors and their parents. Clin Psychol Rev. 2006 May;26(3):233-56. doi: 10.1016/j.cpr.2005.10.002. Epub 2006 Jan 18. PMID 16412542
- [Background] Daviss WB, Mooney D, Racusin R, Ford JD, Fleischer A, McHugo GJ. Predicting posttraumatic stress after hospitalization for pediatric injury. J Am Acad Child Adolesc Psychiatry. 2000 May;39(5):576-83. doi: 10.1097/00004583-200005000-00011. PMID 10802975
- [Background] Farley LM, DeMaso DR, D'Angelo E, Kinnamon C, Bastardi H, Hill CE, Blume ED, Logan DE. Parenting stress and parental post-traumatic stress disorder in families after pediatric heart transplantation. J Heart Lung Transplant. 2007 Feb;26(2):120-6. doi: 10.1016/j.healun.2006.11.013. PMID 17258144
- [Background] Kazak AE, Alderfer M, Rourke MT, Simms S, Streisand R, Grossman JR. Posttraumatic stress disorder (PTSD) and posttraumatic stress symptoms (PTSS) in families of adolescent childhood cancer survivors. J Pediatr Psychol. 2004 Apr-May;29(3):211-9. doi: 10.1093/jpepsy/jsh022. PMID 15131138
- [Background] Shemesh E, Lurie S, Stuber ML, Emre S, Patel Y, Vohra P, Aromando M, Shneider BL. A pilot study of posttraumatic stress and nonadherence in pediatric liver transplant recipients. Pediatrics. 2000 Feb;105(2):E29. doi: 10.1542/peds.105.2.e29. PMID 10654989
- [Background] Stuber ML, Meeske KA, Krull KR, Leisenring W, Stratton K, Kazak AE, Huber M, Zebrack B, Uijtdehaage SH, Mertens AC, Robison LL, Zeltzer LK. Prevalence and predictors of posttraumatic stress disorder in adult survivors of childhood cancer. Pediatrics. 2010 May;125(5):e1124-34. doi: 10.1542/peds.2009-2308. PMID 20435702
- [Background] Landolt MA, Vollrath M, Ribi K, Gnehm HE, Sennhauser FH. Incidence and associations of parental and child posttraumatic stress symptoms in pediatric patients. J Child Psychol Psychiatry. 2003 Nov;44(8):1199-207. doi: 10.1111/1469-7610.00201. PMID 14626460
- [Background] Landolt MA, Ystrom E, Sennhauser FH, Gnehm HE, Vollrath ME. The mutual prospective influence of child and parental post-traumatic stress symptoms in pediatric patients. J Child Psychol Psychiatry. 2012 Jul;53(7):767-74. doi: 10.1111/j.1469-7610.2011.02520.x. Epub 2011 Dec 29. PMID 22211718
- [Background] Bandura A. Self-Efficacy: The Exercise of Control. New York: W.H. Freeman; 1997.
- [Background] Bernstein CM, Stockwell MS, Gallagher MP, Rosenthal SL, Soren K. Mental health issues in adolescents and young adults with type 1 diabetes: prevalence and impact on glycemic control. Clin Pediatr (Phila). 2013 Jan;52(1):10-5. doi: 10.1177/0009922812459950. Epub 2012 Sep 17. PMID 22988007
- [Background] Kakleas K, Kandyla B, Karayianni C, Karavanaki K. Psychosocial problems in adolescents with type 1 diabetes mellitus. Diabetes Metab. 2009 Nov;35(5):339-50. doi: 10.1016/j.diabet.2009.05.002. Epub 2009 Aug 22. PMID 19700362
- [Background] Grossman HY, Brink S, Hauser ST. Self-efficacy in adolescent girls and boys with insulin-dependent diabetes mellitus. Diabetes Care. 1987 May-Jun;10(3):324-9. doi: 10.2337/diacare.10.3.324. PMID 3595399
- [Background] Griva, K., Myers, L.B., & Newman, S. (2000). Illness perceptions and self-efficacy beliefs in adolescents and young adults with insulin dependent diabetes mellitus. Psychology & Health, 15, 733-750.
- [Background] Ott, J., Greening, L., Palardy, N.,… et al. (2000). Self-efficacy as a mediator variable for adolescents' adherence to treatment for insulin-dependent diabetes mellitus. Child Health Care, 29, 47-63.
- [Background] Iannotti RJ, Schneider S, Nansel TR, Haynie DL, Plotnick LP, Clark LM, Sobel DO, Simons-Morton B. Self-efficacy, outcome expectations, and diabetes self-management in adolescents with type 1 diabetes. J Dev Behav Pediatr. 2006 Apr;27(2):98-105. doi: 10.1097/00004703-200604000-00003. PMID 16682872
- [Background] Anderson BJ, Vangsness L, Connell A, Butler D, Goebel-Fabbri A, Laffel LM. Family conflict, adherence, and glycaemic control in youth with short duration Type 1 diabetes. Diabet Med. 2002 Aug;19(8):635-42. doi: 10.1046/j.1464-5491.2002.00752.x. PMID 12147143
- [Background] Palmer DL, Osborn P, King PS, Berg CA, Butler J, Butner J, Horton D, Wiebe DJ. The structure of parental involvement and relations to disease management for youth with type 1 diabetes. J Pediatr Psychol. 2011 Jun;36(5):596-605. doi: 10.1093/jpepsy/jsq019. Epub 2010 Apr 1. PMID 20360016
- [Background] Anderson BJ, Brackett J, Ho J, Laffel LM. An office-based intervention to maintain parent-adolescent teamwork in diabetes management. Impact on parent involvement, family conflict, and subsequent glycemic control. Diabetes Care. 1999 May;22(5):713-21. doi: 10.2337/diacare.22.5.713. PMID 10332671
- [Background] Sheeber L, Hops H, Davis B. Family processes in adolescent depression. Clin Child Fam Psychol Rev. 2001 Mar;4(1):19-35. doi: 10.1023/a:1009524626436. PMID 11388562
- [Background] Wiebe DJ, Berg CA, Korbel C, Palmer DL, Beveridge RM, Upchurch R, Lindsay R, Swinyard MT, Donaldson DL. Children's appraisals of maternal involvement in coping with diabetes: enhancing our understanding of adherence, metabolic control, and quality of life across adolescence. J Pediatr Psychol. 2005 Mar;30(2):167-78. doi: 10.1093/jpepsy/jsi004. PMID 15681311
- [Background] Wysocki T, Taylor A, Hough BS, Linscheid TR, Yeates KO, Naglieri JA. Deviation from developmentally appropriate self-care autonomy. Association with diabetes outcomes. Diabetes Care. 1996 Feb;19(2):119-25. doi: 10.2337/diacare.19.2.119. PMID 8718430
- [Background] Davis CL, Delamater AM, Shaw KH, La Greca AM, Eidson MS, Perez-Rodriguez JE, Nemery R. Parenting styles, regimen adherence, and glycemic control in 4- to 10-year-old children with diabetes. J Pediatr Psychol. 2001 Mar;26(2):123-9. doi: 10.1093/jpepsy/26.2.123. PMID 11181888
- [Background] Butler JM, Skinner M, Gelfand D, Berg CA, Wiebe DJ. Maternal parenting style and adjustment in adolescents with type I diabetes. J Pediatr Psychol. 2007 Nov-Dec;32(10):1227-37. doi: 10.1093/jpepsy/jsm065. Epub 2007 Aug 23. PMID 17717004
- [Background] Baumrind, D. (1971). Current patterns of parental authority. Developmental Psychology, 4(1p2), 1.
- [Background] Baumrind, D. (1966). Effects of authoritative parental control on child behavior. Child Development, 887-907.
- [Background] Darling, N., & Steinberg, L. (1993). Parenting style as context: An integrative model. Psychological bulletin, 113(3), 487.
- [Background] Greene MS, Mandleco B, Roper SO, Marshall ES, Dyches T. Metabolic control, self-care behaviors, and parenting in adolescents with type 1 diabetes: a correlational study. Diabetes Educ. 2010 Mar-Apr;36(2):326-36. doi: 10.1177/0145721710361270. Epub 2010 Mar 3. PMID 20200283
- [Background] Shorer M, David R, Schoenberg-Taz M, Levavi-Lavi I, Phillip M, Meyerovitch J. Role of parenting style in achieving metabolic control in adolescents with type 1 diabetes. Diabetes Care. 2011 Aug;34(8):1735-7. doi: 10.2337/dc10-1602. PMID 21788643
- [Background] Aunola K, Nurmi JE. The role of parenting styles in children's problem behavior. Child Dev. 2005 Nov-Dec;76(6):1144-59. doi: 10.1111/j.1467-8624.2005.00841.x. PMID 16274431
- [Background] Berg CA, Wiebe DJ, Beveridge RM, Palmer DL, Korbel CD, Upchurch R, Swinyard MT, Lindsay R, Donaldson DL. Mother child appraised involvement in coping with diabetes stressors and emotional adjustment. J Pediatr Psychol. 2007 Sep;32(8):995-1005. doi: 10.1093/jpepsy/jsm043. Epub 2007 Jun 14. PMID 17569712
- [Background] Cyranowski JM, Frank E, Young E, Shear MK. Adolescent onset of the gender difference in lifetime rates of major depression: a theoretical model. Arch Gen Psychiatry. 2000 Jan;57(1):21-7. doi: 10.1001/archpsyc.57.1.21. PMID 10632229
- [Background] Oldehinkel AJ, Veenstra R, Ormel J, de Winter AF, Verhulst FC. Temperament, parenting, and depressive symptoms in a population sample of preadolescents. J Child Psychol Psychiatry. 2006 Jul;47(7):684-95. doi: 10.1111/j.1469-7610.2005.01535.x. PMID 16790003
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Birmaher B, Khetarpal S, Brent D, Cully M, Balach L, Kaufman J, Neer SM. The Screen for Child Anxiety Related Emotional Disorders (SCARED): scale construction and psychometric characteristics. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):545-53. doi: 10.1097/00004583-199704000-00018. PMID 9100430
- [Background] Pynoos RS, Frederick C, Nader K, Arroyo W, Steinberg A, Eth S, Nunez F, Fairbanks L. Life threat and posttraumatic stress in school-age children. Arch Gen Psychiatry. 1987 Dec;44(12):1057-63. doi: 10.1001/archpsyc.1987.01800240031005. PMID 3689093
- [Background] Steinberg AM, Brymer MJ, Decker KB, Pynoos RS. The University of California at Los Angeles Post-traumatic Stress Disorder Reaction Index. Curr Psychiatry Rep. 2004 Apr;6(2):96-100. doi: 10.1007/s11920-004-0048-2. PMID 15038911
- [Background] Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. 2007 Jul;164(7):1035-43. doi: 10.1176/ajp.2007.164.7.1035. PMID 17606655
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] . Robinson, C. C., Mandleco, B., Olsen, S. F., & Hart, C. H. (2001). The parenting styles and dimensions questionnaire (PSDQ). Handbook of Family Measurement Techniques, 3, 319-321.
- [Background] Robinson, C. C., Mandleco, B., Olsen, S. F., & Hart, C. H. (1995). Authoritative, authoritarian, and permissive parenting practices: Development of a new measure. Psychological Reports, 77(3), 819-830.